CLINICAL TRIAL: NCT00001217
Title: Osteosarcoma Study #2: A Randomized Trial of Pre-Surgical Chemotherapy vs. Immediate Surgery and Adjuvant Chemotherapy in the Treatment of Non-Metastatic Osteosarcoma. A Pediatric Oncology Group Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 870068; 87-C-0068
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Osteosarcoma
Keywords: Non-Metastatic Osteosarcoma; Presurgical Chemotherapy
MeSH Terms: conditions — Osteosarcoma

INTERVENTIONS:
Drug: pre-surgical chemotherapy

SUMMARY:
The study is designed to determine if the administration of multi-drug adjuvant chemotherapy for patients with primary non-metastatic osteogenic sarcoma, both prior to and after the definitive surgical procedure for their primary tumor is superior as a treatment strategy to the current approach of giving drugs only after the definitive surgical procedure has been performed. An effort will be made as well to determine if the administration of pre-definitive surgery, chemotherapy leads to an increase in the proportion of the patients suitable for a limb salvage primary surgical procedure.

DETAILED DESCRIPTION:
The study is designed to determine if the administration of multi-drug adjuvant chemotherapy for patients with primary non-metastatic osteogenic sarcoma, both prior to and after the definitive surgical procedure for their primary tumor is superior as a treatment strategy to the current approach of giving drugs only after the definitive surgical procedure has been performed. An effort will be made as well to determine if the administration of pre-definitive surgery, chemotherapy leads to an increase in the proportion of the patients suitable for a limb salvage primary surgical procedure.

ELIGIBILITY:
Must be less than or equal to 30 years of age.

No prior history of cancer.

No prior therapy-other than biopsy.

Informed consent according or institutional guidelines (Agreement to randomization to either presurgical chemotherapy or immediate surgery-physicians must also agree).

Less than or equal to 21 days since initial diagnosis and eligible to have surgery within 3 weeks of randomization.

Must have a high grade osteosarcoma.

Must not have low grade osteosarcoma, periosteal and parosteal

osteosarcoma, or multi-focal sclerosing of osteosarcoma.

Tumor must be confined to extremity or expendable and resectable bone of axial skeleton (i.e., ilium, scapula, clavicle, rib).

No evidence of metastases by PE, CXR, chest CT, and bone scans. (Chest CT must be normal within 2 weeks of randomization). Abnormalities on chest CT must be biopsy-negative or thoracotomy negative. Suspicious lesions on bone scan should be biopsied.

LDH level and surgical intent (i.e., amputation, resection, or limb replacement) must be known before patient is registered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260
Dates: Start 1987-05; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosen G, Caparros B, Huvos AG, Kosloff C, Nirenberg A, Cacavio A, Marcove RC, Lane JM, Mehta B, Urban C. Preoperative chemotherapy for osteogenic sarcoma: selection of postoperative adjuvant chemotherapy based on the response of the primary tumor to preoperative chemotherapy. Cancer. 1982 Mar 15;49(6):1221-30. doi: 10.1002/1097-0142(19820315)49:63.0.co;2-e. PMID 6174200
- [Background] Winkler K, Beron G, Kotz R, Salzer-Kuntschik M, Beck J, Beck W, Brandeis W, Ebell W, Erttmann R, Gobel U, et al. Neoadjuvant chemotherapy for osteogenic sarcoma: results of a Cooperative German/Austrian study. J Clin Oncol. 1984 Jun;2(6):617-24. doi: 10.1200/JCO.1984.2.6.617. PMID 6202851
- [Background] Link MP, Goorin AM, Miser AW, Green AA, Pratt CB, Belasco JB, Pritchard J, Malpas JS, Baker AR, Kirkpatrick JA, et al. The effect of adjuvant chemotherapy on relapse-free survival in patients with osteosarcoma of the extremity. N Engl J Med. 1986 Jun 19;314(25):1600-6. doi: 10.1056/NEJM198606193142502. PMID 3520317